CLINICAL TRIAL: NCT01730742
Title: The Role of Sleep Deprivation in the Regulation of Immune System, Neuroendocrine Responses, and Behavioral Measures.
Brief Title: Sleep Deprivation's Regulation of Immune System Function and Behavior
Acronym: SS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 192837465
Record Dates: First submitted 2012-10-11; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Sleep Deprivation; Sleep
MeSH Terms: conditions — Sleep Deprivation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep deprivation (Experimental): Total sleep deprivation: participants were required to stay up for the entire night before a 'Blood Sample' was taken and the 'Neuroeconomics task' and 'Portion size task' were performed
  Interventions: Behavioral: Neuroeconomics task; Behavioral: Portion Size Task; Procedure: Blood sample
- Sleep (Experimental): Sleep: participants had an 8-h sleep opportunity before a 'Blood Sample' was taken and the 'Neuroeconomics task' and 'Portion size task' were performed
  Interventions: Behavioral: Neuroeconomics task; Behavioral: Portion Size Task; Procedure: Blood sample

INTERVENTIONS:
Behavioral: Neuroeconomics task — After a night of wakefulness, participants performed the neuroeconomics task (shopping food items in a mock supermarket scenario).
Behavioral: Portion Size Task — Participants are given a computer program that gives them the opportunity to choose the portions of a variety of food items that they would ideally like to consume
Procedure: Blood sample — After a night of wakefulness, a blood sample was taken to assess the level and efficacy of circulating neutrophils, as well as to assay blood serum and plasma for the presence of hormones involved in hunger such as oxytocin and ghrelin

SUMMARY:
The study proposes to investigate whether sleep deprivation will affect a variety of measures, including hormones, immune system functioning, and behaviors related to food intake and hunger. It is predicted that sleep deprivation will affect circulating neutrophil activity, and do so via affects on DNA methylation. It is also predicted that sleep deprivation will up-regulate ghrelin, and down-regulate circulating oxytocin. Finally, it is predicted that sleep deprivation will increase participants' tendencies to pick larger portions of food, and also increase their tendency to purchase foods that are more caloric in a mock supermarket scenario.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-35y
* Healthy (self-reported) and not on medication
* Non-smoking
* Normal sleep-wake rhythm (i.e. 7-8 h per night, self-reported)

Exclusion Criteria:

* Major illness
* Taking any serious medications
* Any sleep conditions (e.g. irregular bedtimes, sleep complaints)
* Any dietary issues with the food items provided
* A history of endocrine or psychiatric disorders

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Neutrophil phagocytotic function production | Change in 4 neutrophil phagocytotic function from baseline to 36hours later (after the nighttime intervention)
  This project is designed to test the inflammatory capacity of circulating neutrophils. It also aims to investigate if any changes in neutrophil efficacy are governed by alterations in DNA methylation.
  Measured during 36 hours (at 1930 day 1, 0730 and 1930 day 2, 0730 day 3)

SECONDARY OUTCOMES:
Portion Size Task | Change in selected portion size from baseline to 1 hr after consuming a caloric preload
  Participants will be evaluated on their tendency to choose larger or smaller portions of a variety of meal items on a computer screen. This will be conducted both following sleep deprivation and sleep, and changes over the hour will be compared between these conditions.
Neuro-economics task | Change in purchasing behaviour 1 hr after consuming a caloric preload
  Participants will be evaluated on their purchasing behavior with regards to high-calorie and low-calorie food items in a mock supermarket scenario following sleep and sleep deprivation.
Circulating hormone levels | Change in circulating hormone levels from baseline (ie. 1930 - before sleep intervention) to 12hr later (0730 after the nighttime intervention)
  Participants will have their circulating hormone levels taken and analyzed, including ghrelin and oxytocin, to determine if sleep deprivation alters hormone levels related primarily to obesity or weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Christian Benedict, PhD, Principal Investigator — dept. of Neuroscience, Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Nilsson EK, Ernst B, Voisin S, Almen MS, Benedict C, Mwinyi J, Fredriksson R, Schultes B, Schioth HB. Roux-en Y gastric bypass surgery induces genome-wide promoter-specific changes in DNA methylation in whole blood of obese patients. PLoS One. 2015 Feb 24;10(2):e0115186. doi: 10.1371/journal.pone.0115186. eCollection 2015. PMID 25710379
- [Derived] Hogenkamp PS, Nilsson E, Nilsson VC, Chapman CD, Vogel H, Lundberg LS, Zarei S, Cedernaes J, Rangtell FH, Broman JE, Dickson SL, Brunstrom JM, Benedict C, Schioth HB. Acute sleep deprivation increases portion size and affects food choice in young men. Psychoneuroendocrinology. 2013 Sep;38(9):1668-74. doi: 10.1016/j.psyneuen.2013.01.012. Epub 2013 Feb 18. PMID 23428257